CLINICAL TRIAL: NCT06048575
Title: Characteristics of the Attention Provided to Patients With Cholecystitis in Villavicencio Hospitals, Colombia: A Retrospective Cross-sectional Trial.
Brief Title: Cholecystitis in Villavicencio Hospitals
Status: Completed | Type: Observational
Sponsor: Hospital Departamental de Villavicencio (Other)
Collaborators: Cooperative University of Colombia (Other)
Responsible Party: Principal Investigator, Norton Perez-Gutierrez, MD, Principal investigator, Hospital Departamental de Villavicencio
Other Study IDs: GRIVI_2023_04_Cholecystitis
Record Dates: First submitted 2023-09-16; First posted 2023-09-21 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Biliary Tract Diseases
Keywords: Acute Cholecystitis; Gallbladder Diseases; Cholecystolithiasis; Biliary Tract Surgical Procedures; Laparoscopy; Conversion to Open Surgery; Hospital Surgery Department; Colombia
MeSH Terms: conditions — Biliary Tract Diseases; Cholecystitis, Acute; Gallbladder Diseases; Cholecystolithiasis | interventions — Cholecystectomy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Number of patients with early therapy: Patients with early surgery (<72 hours of admission).
  Interventions: Procedure: Cholecystectomy
- Number of patients with subacute therapy: Patients with surgery for three days or more.
  Interventions: Procedure: Cholecystectomy
- Number of patients with late therapy: Patients with surgery beyond ten days.
  Interventions: Procedure: Cholecystectomy
- Number of patients with no therapy: Patients discharged with no surgical therapy.
  Interventions: Procedure: Cholecystectomy

INTERVENTIONS:
Procedure: Cholecystectomy — Early or late surgery, ambulatory, emergency, or differed.

SUMMARY:
Background: Acute cholecystitis is a frequent cause of visits to the emergency ward. The complications of delays in attention and surgical therapy are substantial and should be considered to prevent them timely.

Objective: The study aims to evaluate the assistance provided to patients for cholecystitis in Villavicencio hospitals.

Methodology: A retrospective cross-sectional trial will be performed. The source of information will be the surgical database of hospitals at Villavicencio from 2019 to 2022. The records selected will be exported to an Excel spreadsheet for debugging and analysis. The central distribution and dispersion of numerical variables will be analyzed, as frequency and proportion of categorical variables with the software Prism 10.01.1 for Mac iOS. Chi-square and U-Mann & Whitney tests will compare variables according to the data type. A p<0.05 will be defined as statistically significant.

Expected results: the researchers hope to define the frequency of hospital discharges due to acute cholecystitis, the type of procedure performed, complications, and outcomes.

Conclusions: The research is feasible because the necessary information is available for evaluation, and it is helpful for the institutions and the region.

DETAILED DESCRIPTION:
Biliary diseases are some leading causes of admission to emergency wards. Cholelithiasis and acute cholecystitis are prevalent in the Orinoquia region. Young and female populations are predominantly affected. Complications are prone to delayed definitive surgical therapy, which increases costs and the use of resources. Guidelines recommend early surgery during hospitalization for the first episode to minimize difficulties. There are limitations in the available technology recommended for treatment, especially in institutions dedicated to vulnerable populations. Laparoscopic cholecystectomy is the primary goal in cases required for gall bladder removal. Although the technology and trained personnel are available in local institutions, open procedures are still performed primarily, and restrictions are due to insurance coverage after more than 30 years of disseminating laparoscopic cholecystectomy worldwide.

It is necessary to know the prevalence of the disease and the therapy provided in general hospitals from the region to analyze associated factors with undesired results.

Determining the characteristics of patients admitted to hospitals by biliary pathology will provide essential information on the severity, care provided, definitive treatment, opportunity, and outcomes. Such an analysis will give knowledge to prioritize policies and resources, upgrade clinical practice guidelines, and improve early and long-term results.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted with acute or chronic biliary pathology.

Exclusion Criteria:

* None.

Ages: 16 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The trial participants are those admitted requesting emergency, hospital, ambulatory, or ICU attention for biliary pathology during the study period, according to the admission registers.
Sampling Method: Non-Probability Sample
Enrollment: 609 (Actual)
Dates: Start 2025-08-01 (Actual); Primary Completion 2025-10-31 (Actual); Study Completion 2025-10-31 (Actual)

PRIMARY OUTCOMES:
Mortality | 28 days
  Number of patients deceased due to the biliary disease, complications, or other conditions.

SECONDARY OUTCOMES:
Hospital length of stay | 28 days
  Number of days before discharge.
Need of ICU | 28 days
  Patients admitted to ICU under any circumstance.
ICU length of stay | 28 days
  Number of days hospitalized in ICU
Surgical site infection | 28 days
  Number of patients with infections associated with the procedure (superficial, deep, organ/space)
Need of mechanical ventilation | 28 days
  Number of patients needing mechanical ventilation
Complicated presentation | 28 days
  Number of patients with complications of the disease previous or during hospitalization, but not related to the surgical procedure
Surgical complications | 28 days
  Number of patients with complications related to the surgical procedure

CONTACTS AND LOCATIONS:
Overall Officials: Norton Perez, MD, Principal Investigator — Cooperative University of Colombia
Locations (1):
- Clinica Primavera, Villavicencio, Meta Department, Colombia

IPD SHARING:
Plan to Share IPD: Undecided
According to the decision of the ethical committee, the database might be stored in the repository of the university.

REFERENCES:
- [Result] Serna JC, Patiño S, Buriticá M, Osorio E, Morales CH, Toro JP. Incidencia de lesión de vías biliares en un hospital universitario: análisis de más de 1.600 colecistectomías laparoscópicas. Rev Colomb Cir. 2019;34(1):45-54.
- [Result] Sanchez Beorlegui J, Monsalve Laguna E, Aspiroz Sancho A, Moreno de Marcos N. Colecistectomía laparoscópica en octogenarios. Rev Colomb Cir. 2008;23(3):136-45.
- [Result] Castro F, Galindo J, Bejarano M. Complicaciones de colecistitis aguda en pacientes operados de urgencia. Rev Colomb Cir. 2008;23(1):15-21.
- [Result] Domínguez LC, Herrera WE, Rivera AM, Bermúdez CE. Colecistectomía de urgencia por laparoscopia por colecistitis aguda en adultos mayores. Rev Colomb Cir. 2011;26:93-100.
- [Result] Díaz S, Correa MJ, Giraldo LM, Ríos DC, Solórzano F, Wolff JD, et al. Experiencia en colecistectomía por laparoscopia en la Clínica Universitaria CES. Rev Colomb Cir. 2012;27(4):275-80.
- [Result] Gaitán JA, Martínez VM. Enfermedad litiásica biliar, experiencia en una clínica de cuarto nivel, 2005-2011. Rev Colomb Cir. 2014;29(3):188-96.
- [Result] Salinas C, López CA, Ramírez A, Torres R, Mendoza MC, Cuesta DP, et al. Colecistectomía por laparoscopia en colecistitis subaguda: análisis retrospectivo de pacientes en un hospital universitario. Rev Colomb Cir. 2018;33(2):154-61.
- [Result] Ángel-González MS, Díaz-Quintero CA, Aristizábal-Arjona F, Turizo-Agamez Á, Molina-Céspedes I, Velásquez-Martínez MA, et al. Controversias en el manejo de la colecistitis aguda tardía. Rev Colomb Cir. 2019;34(4):364-71.
- [Result] Arroyave Y, Torres F, Sarzosa F, Díaz J, Arroyave Y, Torres F, et al. ¿Es más difícil la colecistectomía laparoscópica después de una colangiopancreatografía retrógrada endoscópica? Experiencia en un hospital de tercer nivel. Rev Colomb Cir. 2020;35(3):436-48.
- [Result] Bustos-Guerrero AM, Guerrero-Macías SI, Manrique-Hernández EF, Gomez-Rincón GA. Severidad de la colecistitis aguda en tiempos de COVID-19: ¿mito o realidad? Rev Colomb Cir. 2022;37(2):206-13.
- [Result] Vargas Rodríguez LJ, Agudelo Sanabria MB, Lizcano Contreras RA, Martínez Balaguera YM, Velandia Bustcara EL, Sánchez Hernández SJ, et al. Factores asociados con la conversión de la colecistectomía laparoscópica a colecistectomía abierta. Rev Colomb Gastroenterol. 2017;32(1):20-3.
- [Result] Yurgaky-Sarmiento J, Otero-Regino W, Gómez-Zuleta M, Yurgaky-Sarmiento J, Otero-Regino W, Gómez-Zuleta M. Elevación de las aminotransferasas: una nueva herramienta para el diagnóstico de coledocolitiasis. Un estudio de casos y controles. Rev Colomb Gastroenterol. 2020;35(3):319-28.
- [Result] Toro-Calle J, Guzmán-Arango C, Ramírez-Ceballos M, Guzmán-Arango N, Toro-Calle J, Guzmán-Arango C, et al. ¿Son los criterios de la ASGE suficientes para la estratificación del riesgo de coledocolitiasis? Rev Colomb Gastroenterol. 2020;35(3):304-10.
- [Result] Busto Bea V, Caro Paton A, Aller Dela Fuente R, Gonzalez Sagrado M, Garcia-Alonso FJ, Perez-Miranda Castillo M. Acute calculous cholecystitis: a real-life management study in a tertiary teaching hospital. Rev Esp Enferm Dig. 2019 Sep;111(9):667-671. doi: 10.17235/reed.2019.6260/2019. PMID 31317760
- [Result] Janikow C, Corti E, Menso N, Moretti G, Ale M, Sanchez M, Lada PE. Useful of Tokyo guidelines in the diagnosis of acute cholecystitis. Anatomopathologie correlationship. Rev Fac Cien Med Univ Nac Cordoba. 2017;74(2):88-92. PMID 28657526
- [Result] Ongen G, Nas OF, Aksoy F, Candan S, Dundar HZ, Ozpar R, Inecikli MF, Gursel BE, Tasar P, Savci G. Comparison of severity and complication rates of acute cholecystitis during pandemic and pre-pandemic periods? Acta Radiol. 2023 Apr;64(4):1363-1370. doi: 10.1177/02841851221137048. Epub 2022 Nov 22. PMID 36412110
- [Result] Lacka M, Obloj P, Spychalski P, Laski D, Rostkowska O, Wieszczy P, Kobiela J. Clinical presentation and outcomes of cholecystectomy for acute cholecystitis in patients with diabetes - A matched pair analysis. A pilot study. Adv Med Sci. 2020 Sep;65(2):409-414. doi: 10.1016/j.advms.2020.08.001. Epub 2020 Aug 18. PMID 32823170
- [Result] Rodriguez-Sanjuan JC, Arruabarrena A, Sanchez-Moreno L, Gonzalez-Sanchez F, Herrera LA, Gomez-Fleitas M. Acute cholecystitis in high surgical risk patients: percutaneous cholecystostomy or emergency cholecystectomy? Am J Surg. 2012 Jul;204(1):54-9. doi: 10.1016/j.amjsurg.2011.05.013. Epub 2011 Oct 13. PMID 22000114
- [Result] Simorov A, Ranade A, Parcells J, Shaligram A, Shostrom V, Boilesen E, Goede M, Oleynikov D. Emergent cholecystostomy is superior to open cholecystectomy in extremely ill patients with acalculous cholecystitis: a large multicenter outcome study. Am J Surg. 2013 Dec;206(6):935-40; discussion 940-1. doi: 10.1016/j.amjsurg.2013.08.019. Epub 2013 Oct 8. PMID 24112675
- [Result] Bourikian S, Anand RJ, Aboutanos M, Wolfe LG, Ferrada P. Risk factors for acute gangrenous cholecystitis in emergency general surgery patients. Am J Surg. 2015 Oct;210(4):730-3. doi: 10.1016/j.amjsurg.2015.05.003. Epub 2015 Jun 27. PMID 26186803
- [Result] Madni TD, Leshikar DE, Minshall CT, Nakonezny PA, Cornelius CC, Imran JB, Clark AT, Williams BH, Eastman AL, Minei JP, Phelan HA, Cripps MW. The Parkland grading scale for cholecystitis. Am J Surg. 2018 Apr;215(4):625-630. doi: 10.1016/j.amjsurg.2017.05.017. Epub 2017 Jun 6. PMID 28619262
- [Result] Lee W, Jang JY, Cho JK, Hong SC, Jeong CY. Does surgical difficulty relate to severity of acute cholecystitis? Validation of the parkland grading scale based on intraoperative findings. Am J Surg. 2020 Apr;219(4):637-641. doi: 10.1016/j.amjsurg.2018.12.005. Epub 2018 Dec 8. PMID 31718816
- [Result] Choi SB, Han HJ, Kim CY, Kim WB, Song TJ, Suh SO, Kim YC, Choi SY. Early laparoscopic cholecystectomy is the appropriate management for acute gangrenous cholecystitis. Am Surg. 2011 Apr;77(4):401-6. PMID 21679545
- [Result] Caputo P, Rossi G, Faccini M, Carzaniga P. Overcoming of a "surgical dogma" in acute cholecystitis treated in postponed emergency. Ann Ital Chir. 2009 Jul-Aug;80(4):287-92. PMID 19967887
- [Result] Clavien PA, Strasberg SM. Severity grading of surgical complications. Ann Surg. 2009 Aug;250(2):197-8. doi: 10.1097/SLA.0b013e3181b6dcab. No abstract available. PMID 19638901
- [Result] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542
- [Result] Gutt CN, Encke J, Koninger J, Harnoss JC, Weigand K, Kipfmuller K, Schunter O, Gotze T, Golling MT, Menges M, Klar E, Feilhauer K, Zoller WG, Ridwelski K, Ackmann S, Baron A, Schon MR, Seitz HK, Daniel D, Stremmel W, Buchler MW. Acute cholecystitis: early versus delayed cholecystectomy, a multicenter randomized trial (ACDC study, NCT00447304). Ann Surg. 2013 Sep;258(3):385-93. doi: 10.1097/SLA.0b013e3182a1599b. PMID 24022431
- [Result] Cooper S, Donovan M, Grieve DA. Outcomes of percutaneous cholecystostomy and predictors of subsequent cholecystectomy. ANZ J Surg. 2018 Jul-Aug;88(7-8):E598-E601. doi: 10.1111/ans.14251. Epub 2017 Oct 20. PMID 29052940
- [Result] Chen H, Jorissen R, Walcott J, Nikfarjam M. Incidence and predictors of common bile duct stones in patients with acute cholecystitis: a systematic literature review and meta-analysis. ANZ J Surg. 2020 Sep;90(9):1598-1603. doi: 10.1111/ans.15565. Epub 2019 Nov 19. PMID 31743951
- [Result] Abi-Haidar Y, Sanchez V, Williams SA, Itani KM. Revisiting percutaneous cholecystostomy for acute cholecystitis based on a 10-year experience. Arch Surg. 2012 May;147(5):416-22. doi: 10.1001/archsurg.2012.135. PMID 22785633
- [Result] Felicio SJO, Matos EP, Cerqueira AM, Farias KWSF, Silva RA, Torres MO. MORTALITY OF URGENCY VERSUS ELECTIVE VIDEOLAPAROSCOPIC CHOLECYSTECTOMY FOR ACUTE CHOLECYSTITIS. Arq Bras Cir Dig. 2017 Jan-Mar;30(1):47-50. doi: 10.1590/0102-6720201700010013. PMID 28489169
- [Result] Wang L, Yu HF, Guo T, Xie P, Zhang ZW, Yu YH. Early Versus Delayed Laparoscopic Cholecystectomy for Acute Cholecystitis with Mild Pancreatitis. Curr Med Sci. 2020 Oct;40(5):937-942. doi: 10.1007/s11596-020-2275-0. Epub 2020 Oct 29. PMID 33123907
- [Result] Dimou FM, Adhikari D, Mehta HB, Riall TS. Outcomes in Older Patients with Grade III Cholecystitis and Cholecystostomy Tube Placement: A Propensity Score Analysis. J Am Coll Surg. 2017 Apr;224(4):502-511.e1. doi: 10.1016/j.jamcollsurg.2016.12.021. Epub 2017 Jan 6. PMID 28069529
- [Result] Nassar AHM, Khan KS, Ng HJ, Sallam M. Operative Difficulty, Morbidity and Mortality Are Unrelated to Obesity in Elective or Emergency Laparoscopic Cholecystectomy and Bile Duct Exploration. J Gastrointest Surg. 2022 Sep;26(9):1863-1872. doi: 10.1007/s11605-022-05344-7. Epub 2022 May 31. PMID 35641812
- [Result] Nasr MM. An Innovative Emergency Laparoscopic Cholecystectomy Technique; Early Results Towards Complication Free Surgery. J Gastrointest Surg. 2017 Feb;21(2):302-311. doi: 10.1007/s11605-016-3308-7. Epub 2016 Oct 25. PMID 27783342
- [Result] Strasberg SM. Avoidance of biliary injury during laparoscopic cholecystectomy. J Hepatobiliary Pancreat Surg. 2002;9(5):543-7. doi: 10.1007/s005340200071. PMID 12541037
- [Result] Miura F, Okamoto K, Takada T, Strasberg SM, Asbun HJ, Pitt HA, Gomi H, Solomkin JS, Schlossberg D, Han HS, Kim MH, Hwang TL, Chen MF, Huang WS, Kiriyama S, Itoi T, Garden OJ, Liau KH, Horiguchi A, Liu KH, Su CH, Gouma DJ, Belli G, Dervenis C, Jagannath P, Chan ACW, Lau WY, Endo I, Suzuki K, Yoon YS, de Santibanes E, Gimenez ME, Jonas E, Singh H, Honda G, Asai K, Mori Y, Wada K, Higuchi R, Watanabe M, Rikiyama T, Sata N, Kano N, Umezawa A, Mukai S, Tokumura H, Hata J, Kozaka K, Iwashita Y, Hibi T, Yokoe M, Kimura T, Kitano S, Inomata M, Hirata K, Sumiyama Y, Inui K, Yamamoto M. Tokyo Guidelines 2018: initial management of acute biliary infection and flowchart for acute cholangitis. J Hepatobiliary Pancreat Sci. 2018 Jan;25(1):31-40. doi: 10.1002/jhbp.509. Epub 2018 Jan 8. PMID 28941329
- [Result] Panni RZ, Chatterjee D, Panni UY, Robbins KJ, Liu J, Strasberg SM. Sequential histologic evolution of gallbladder inflammation in acute cholecystitis over the first 10 days after onset of symptoms. J Hepatobiliary Pancreat Sci. 2023 Jun;30(6):724-736. doi: 10.1002/jhbp.1274. Epub 2022 Dec 1. PMID 36399043
- [Result] Yokoe M, Takada T, Strasberg SM, Solomkin JS, Mayumi T, Gomi H, Pitt HA, Gouma DJ, Garden OJ, Buchler MW, Kiriyama S, Kimura Y, Tsuyuguchi T, Itoi T, Yoshida M, Miura F, Yamashita Y, Okamoto K, Gabata T, Hata J, Higuchi R, Windsor JA, Bornman PC, Fan ST, Singh H, de Santibanes E, Kusachi S, Murata A, Chen XP, Jagannath P, Lee S, Padbury R, Chen MF; Tokyo Guidelines Revision Committee. New diagnostic criteria and severity assessment of acute cholecystitis in revised Tokyo Guidelines. J Hepatobiliary Pancreat Sci. 2012 Sep;19(5):578-85. doi: 10.1007/s00534-012-0548-0. PMID 22872303
- [Result] Yokoe M, Takada T, Hwang TL, Endo I, Akazawa K, Miura F, Mayumi T, Mori R, Chen MF, Jan YY, Ker CG, Wang HP, Itoi T, Gomi H, Kiriyama S, Wada K, Yamaue H, Miyazaki M, Yamamoto M. Descriptive review of acute cholecystitis: Japan-Taiwan collaborative epidemiological study. J Hepatobiliary Pancreat Sci. 2017 Jun;24(6):319-328. doi: 10.1002/jhbp.450. Epub 2017 May 14. PMID 28316140
- [Result] Endo I, Takada T, Hwang TL, Akazawa K, Mori R, Miura F, Yokoe M, Itoi T, Gomi H, Chen MF, Jan YY, Ker CG, Wang HP, Kiriyama S, Wada K, Yamaue H, Miyazaki M, Yamamoto M. Optimal treatment strategy for acute cholecystitis based on predictive factors: Japan-Taiwan multicenter cohort study. J Hepatobiliary Pancreat Sci. 2017 Jun;24(6):346-361. doi: 10.1002/jhbp.456. Epub 2017 May 31. PMID 28419741
- [Result] Schuster KM, O'Connor R, Cripps M, Kuhlenschmidt K, Taveras L, Kaafarani HM, El Hechi M, Puri R, Schroeppel TJ, Enniss TM, Cullinane DC, Cullinane LM, Agarwal S Jr, Kaups K, Crandall M, Tominaga G. Revision of the AAST grading scale for acute cholecystitis with comparison to physiologic measures of severity. J Trauma Acute Care Surg. 2022 Apr 1;92(4):664-674. doi: 10.1097/TA.0000000000003507. PMID 34936593
- [Result] Mercado MA. [From Langenbuch to Strasberg: the spectrum of bile duct injuries]. Rev Invest Clin. 2004 Sep-Oct;56(5):649-64. Spanish. PMID 15776870
- [Result] Sugiura R, Nakamura H, Horita S, Meguro T, Sasaki K, Kagaya H, Yoshida T, Aoki H, Morita T, Fujita M, Tamoto E, Fukushima M, Ashitate Y, Ueno T, Tsutaho A, Kuwatani M, Sakamoto N. Assessment of postoperative common bile duct stones after endoscopic extraction and subsequent cholecystectomy. Surg Endosc. 2022 Sep;36(9):6535-6542. doi: 10.1007/s00464-022-09017-z. Epub 2022 Jan 18. PMID 35041052
- [Result] Welsh S, Nassar AHM, Sallam M. The incidence, operative difficulty and outcomes of staged versus index admission laparoscopic cholecystectomy and bile duct exploration for all comers: a review of 5750 patients. Surg Endosc. 2022 Nov;36(11):8221-8230. doi: 10.1007/s00464-022-09272-0. Epub 2022 May 4. PMID 35507063
- [Result] Borzellino G, Sauerland S, Minicozzi AM, Verlato G, Di Pietrantonj C, de Manzoni G, Cordiano C. Laparoscopic cholecystectomy for severe acute cholecystitis. A meta-analysis of results. Surg Endosc. 2008 Jan;22(1):8-15. doi: 10.1007/s00464-007-9511-6. Epub 2007 Aug 18. PMID 17704863
- [Result] Huang SZ, Chen HQ, Liao WX, Zhou WY, Chen JH, Li WC, Zhou H, Liu B, Hu KP. Comparison of emergency cholecystectomy and delayed cholecystectomy after percutaneous transhepatic gallbladder drainage in patients with acute cholecystitis: a systematic review and meta-analysis. Updates Surg. 2021 Apr;73(2):481-494. doi: 10.1007/s13304-020-00894-4. Epub 2020 Oct 13. PMID 33048340
- [Result] Derici H, Kara C, Bozdag AD, Nazli O, Tansug T, Akca E. Diagnosis and treatment of gallbladder perforation. World J Gastroenterol. 2006 Dec 28;12(48):7832-6. doi: 10.3748/wjg.v12.i48.7832. PMID 17203529